CLINICAL TRIAL: NCT02535468
Title: T2Bacteria Panel Pivotal Study
Acronym: T2Bacteria
Status: Completed | Type: Observational
Sponsor: T2 Biosystems (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-00400
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Bacteremia
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prospective Arm
- Contrived Arm

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of the T2Bacteria Panel by validating the clinical performance (i.e. estimated sensitivity and specificity) of the T2Bacteria Panel compared to blood culture results and/or known Bacteria positive status of prospectively collected clinical specimens and contrived (i.e. Bacteria-spiked) whole blood "clinical samples".

ELIGIBILITY:
Inclusion Criteria:

* Subject or subject's legally authorized representative (LAR) must be able to understand, read and sign the study specific informed consent form after the nature of the study has been fully explained to them.
* Subject has had a diagnostic blood culture ordered, per routine standard of care (prospective arm only).
* Subject is between 18-95 years of age.

Exclusion Criteria:

* Subject has other co-morbid condition(s) that, in the opinion of the Investigator, could limit the subject's ability to participate in the study or impact the scientific integrity of the study.
* Subject has had previous specimens tested by the T2Bacteria Panel with valid results.
* Treatment of subject with any investigational novel drug compound within 30 days prior to the collection of T2 specimens.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates participating in the prospective arm of the study will come from the hospital population who have had a blood culture ordered per routine standard of care. The contrived arm of the study is open to any participants that meet the study enrollment criteria. The study population for both arms is defined as all subjects who meet the study eligibility criteria, provide informed consent, and provide the clinical specimens under this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 2430 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity | Up to 19 hours post blood collection
  The primary endpoint of estimated sensitivity will be determined by comparing positive blood culture results with the concomitantly collected T2Bacteria Panel results from the prospective clinical specimens. PPA will estimated based on the positive T2Bacteria detections of contrived clinical samples.
Specificity | Up to 19 hours post blood collection
  The primary endpoint of estimated specificity will be determined by comparing the negative blood culture results with the concomitantly collected T2Bacteria Panel results from the prospective clinical specimens. NPA will be estimated based on the negative contrived clinical samples.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Henry Ford Health System, Detroit, Michigan
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island